CLINICAL TRIAL: NCT05242497
Title: Effectiveness and Safety of Pharmacopuncture Therapy for Patients with Lumbar Spinal Stenosis : Multicentered, Pragmatic Randomized Controlled, Parallel Grouped Study
Brief Title: Effectiveness and Safety of Pharmacopuncture Therapy for Patients with Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-14
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pharmacopuncture group (Experimental): The physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Interventions: Procedure: pharmacopuncture
- conservative treatment group (Active Comparator): The physicians will choose the type and time of physical therapy and if needed, pharmacological treatment according to participants' conditions.
  Interventions: Procedure: conservative treatments (including physiotherapy)

INTERVENTIONS:
Procedure: pharmacopuncture — This is a pragmatic randomized controlled trials, so the physicians will choose pharmacopuncture treatment, including the type and doses, according to each participant's conditions. The researcher will record the specific intervention precisely and concurrently.
  Arms: pharmacopuncture group
Procedure: conservative treatments (including physiotherapy) — This is a pragmatic randomized controlled trials, so the physicians will choose conservative treatment, including physiotherapy and pharmacological treatment, according to each participant's conditions. The researcher will record the specific intervention precisely and concurrently.
  Arms: conservative treatment group

SUMMARY:
This is 1:1 pragmatic randomized controlled trials in a parallel-grouped, multi-centered design that investigated pharmacopuncture therapy for patients with lumbar spinal stenosis, compared to the conservative treatments including physiotherapy and pharmacological treatments.

DETAILED DESCRIPTION:
This is 1:1 pragmatic randomized controlled trials in a parallel-grouped, multi-centered design that investigated pharmacopuncture therapy for patients with lumbar spinal stenosis, compared to the conservative treatments including physiotherapy and pharmacological treatments. The physician will decide specific location, type, and doses of pharmacopuncture therapy or conservative treatments according to each participants' disease conditions, respectively. The researcher will record concurrently.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with lumbar spinal stenosis based on radiology including computed tomography or magnetic resonance imaging.
2. Clear neurogenic claudication symptoms existed (symptoms aggravated with walking, and alleviated upon resting in lumbar flexion position).
3. reported radiating leg pain or low back pain (LBP) with intensity of NRS ≥5
4. Between the age of 19 and 69 years old.
5. Participants who agreed to participate the study and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Patients with vascular claudication
2. Patients with pathologies of non-spinal origin that may cause LBP or radiating leg pain (e.g. spinal tumor, fracture)
3. Patients with soft tissue pathologies that may cause LBP or radiating leg pain (e.g. tumor, fibromyalgia, rheumatoid arthritis, gout)
4. Patients with other systemic diseases that may interfere with treatment effect or outcome interpretation
5. Patients who administrate those prescribed medicine that may interfere with interpretation of the result (e.g. corticosteroids, immunosuppressants, physchotropic drugs)
6. Patients for whom pharmacopuncture treatment may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, serious diabetes with risk of infection)
7. Patients who were treated with one of the following intervention within the past week; medicine that may potentially influence pain such as NSAIDs (nonsteroidal antiinflammatory drugs), pharmacopuncture, or physical therapies.
8. Pregnant patients or patients planning pregnancy
9. Patients with medical history of spinal surgery within the past 3 months
10. Previous participation in other clinical studies within 1 month of current study enrollment, or plans to participate in other clinical studies during participation (including follow-up period) of the current study after study enrollment
11. Patients unable to fill out study participation consent form
12. Patients deemed unsuitable for study participation as assessed by the researchers

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | week 13
  NRS is a pain scale in which the patients indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'. The NRS of major painful site, which was chosen between low back and radiation pain in lower extremities, will be reported.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of low back pain and radiating pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 25, 53
  NRS is a pain scale in which the patients indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual analogue scale (VAS) of low back pain and radiating pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 25, 53
  The patient indicates their pain severity from minimum 0 to maximum 100, which is a higher score means a worse outcome. VAS of low back pain and radiating leg pain will be reported.
Walking distance | week 1, 5, 9, 13, 25, 53
  Claudication-free walking distance and maximal walking distance will be evaluated.
Zurich Claudication Questionnaire (ZCQ) | week 1, 5, 9, 13, 25, 53
  ZCQ is a lumbar spinal stenosis-specific patient reported outcome, which evaluate the disease severity, functional scale and satisfaction at the treatment.
Oswestry disability index (ODI) | week 1, 5, 9, 13, 25, 53
  ODI is a functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome).
PGIC | week 13, 25, 53
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
Short Form-12 Health Survey version 2 (SF-12 v2) | week 1, 5, 9, 13, 25, 53
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | week 1, 5, 9, 13, 25, 53
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, Ph.D, Study Director — Jaseng Medical Foundation
Locations (7):
- South Korea (7):
  - Dongguk University Bundang Oriental Hospital, Seongnam-si, Bundang-gu
  - Kyung Hee University Korean Medicine Hospital, Seoul, Dongdaemun-gu
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul, Gangdong-gu
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Park KS, Kim S, Seo JY, Cho HW, Nam D, Park Y, Kim EJ, Lee YJ, Ha IH. The Effectiveness of Pharmacopuncture in Patients with Lumbar Spinal Stenosis: A Protocol for a Multi-Centered, Pragmatic, Randomized, Controlled, Parallel Group Study. J Pain Res. 2022 Sep 23;15:2989-2996. doi: 10.2147/JPR.S382550. eCollection 2022. PMID 36176963